CLINICAL TRIAL: NCT02881021
Title: Effects of Kinesiotaping Added to a Rehabilitation Program for Patients With Rotator Cuff Tendinopathy: Protocol of a Single-blind Randomized Controlled Trial Addressing Symptoms, Functional Limitations, and Underlying Deficits.
Brief Title: Effects of Kinesiotaping on Symptoms, Functional Limitations, and Underlying Deficits of Patients With Rotator Cuff Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Fabio Oliveira, PT, MSc, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FOliveira
Record Dates: First submitted 2016-08-12; First posted 2016-08-26 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Rotator Cuff Tendinopathy
Keywords: elastic tape; kinesiology taping; physiotherapy; rotator cuff; shoulder pain; tendon injuries
MeSH Terms: conditions — Shoulder Pain; Tendon Injuries | interventions — Rehabilitation; Bandages; Athletic Tape

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rehabilitation program and kinesiotaping. (Experimental): Each patient will attend 10 physiotherapy sessions over six. Patients from the Experimental group (KT group) will receive the same standardized rehabilitation program as control group (No-KT group) including manual therapy, movement training, stretching, muscular strengthening, and patient education.
  Only KT-group (experimental) will receive therapeutic KT added to the rehabilitation program.
  Kinesio® Tex Classic will be applied using a combination of techniques designed for RCTe and underlying symptoms following the instructions and principles described by Kase et al (2003).
  Kinesiotaping strips will be weaned gradually, according to the individual improvements of deficits evaluated weekly by the physiotherapist treating.
  Interventions: Other: Rehabilitation program; Device: Kinesiotaping
- Rehabilitation program. (Active Comparator): Each patient will attend 10 physiotherapy sessions over six. Patients allocated at the control group (No-KT group) will receive only the rehabilitation program, including manual therapy, movement training, stretching, muscular strengthening, and patient education.
  The rehabilitation program will be exactly the same applied to the experimental group (KT group).
  Interventions: Other: Rehabilitation program

INTERVENTIONS:
Other: Rehabilitation program — Standardized conventional evidence-based physiotherapy for treating rotator cuff tendinopathy.
Device: Kinesiotaping — Combined Kinesiotaping techniques (3 strips) for rotator cuff tendinopathy, following the principles of Kenzo Kase et al. (2003).
  Other Names: Kinesio Tex Classic; Elastic tape; bandage; taping; Kinesio Tape; Kinesiology tape; Kinesiotape
  Arms: Rehabilitation program and kinesiotaping.

SUMMARY:
Introduction: Rotator cuff tendinopathy (RCTe) is the most frequent cause of shoulder pain, resulting in considerable losses to society and public resources. Muscle imbalance and inadequate sensorimotor control are deficits often associated with RCTe. Kinesiotaping (KT) is widely used by clinicians for rehabilitation of RCTe. While previous studies have examined the immediate effects of KT on shoulder injuries or the effects of KT as an isolated method of treatment, no published study has addressed its mid- and long-term effects when combined to a rehabilitation program for patients with RCTe. The primary objective of this randomised controlled trial (RCT) will be to assess the efficacy of therapeutic KT, added to a rehabilitation program, in reducing pain and disabilities in individuals with RCTe. Secondary objectives will look at the effects of KT on the underlying factors involved in shoulder control, such as muscular activity, acromiohumeral distance (AHD), and range of motion (ROM).

Methods and analysis: A single-blind RCT will be conducted. Fifty-two participants, randomly allocated to one of two groups (KT or no-KT), will take part in a 6-week rehabilitation program. The KT-group will receive KT added to the rehabilitation program, whereas the no-KT group will receive only the rehabilitation program. Measurements will be taken at baseline, week-3, week-6, week-12 and 6-month. Primary outcomes will be symptoms and functional limitations assessed by the DASH questionnaire. Secondary outcomes will include shoulder ROM, AHD at rest and at 60º of abduction, and muscle activation during arm elevation. The added effects of KT will be assessed through a 2-way ANOVA for repeated measures.

Discussion: Investigations with a high level of evidence are needed to determine scientific evidence-based concerning the efficacy of KT for the rehabilitation of individuals with RCTe. This RCT will be the first to assess the effectiveness of KT added into a conventional RP for patients with RCTe, addressing underlying factors that could explain the possible benefits of this method, in a mid- and long-term. Results may contribute to build solid evidence on the addition of KT in a physiotherapy intervention for this population.

Ethics and Dissemination: Ethics approval was obtained from the Ethics Committee of Quebec Rehabilitation Institute (IRDPQ) of the CIUSS-CN. Results of this protocol will be disseminated through international publications in peer-reviewed journals, in addition to international conference presentations.

ELIGIBILITY:
Inclusion Criteria.

To be eligible, participants should have unilateral rotator cuff tendinopathy and to present one positive finding in each of the following categories:

* Painful arc of movement during flexion or abduction;
* Neer (sensitivity 0.78, specificity 0.58) or Kennedy-Hawkins impingement signs (sensitivity 0.74, specificity 0.57);
* Pain on resisted external rotation, abduction or empty can test (sensitivity 0.69, specificity 0.62).

Exclusion Criteria.

Patients will be excluded if they have:

* an open wound that compromises KT application;
* had a previous shoulder surgery;
* allergy or intolerance to KT;
* adhesive capsulitis, defined as loss of passive shoulder ROM greater than 50%;
* history of glenohumeral luxation or fracture to the shoulder girdle;
* shoulder pain reproduced by cervical movements;
* clinical signs of full-thickness RC tears identified by lag signs tests (drop, internal, and external rotation signs).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
Functional Limitations (changes during treatment; from baseline to 6 months follow-up). | Week-0 (baseline), week-3 (mid-point of the treatment), week-6 (end of treatment), week-12 (mid-term follow-up), 6-month (long-term follow-up).
  Functional limitations will be measured throughout treatment using "The Disabilities of the Arm, Shoulder, and Hand (DASH)".
  The DASH is a 30-item self-report questionnaire, designed to measure physical disability and symptoms of upper limbs disorders. A validated Canadian-French version will be used (Intraclass correlation coefficient (ICC)=0.93; standardized response mean (SRM)=1.35; minimal detectable change (MDC)=11.4 points; clinically important difference (CID)=10 points)
Symptoms (pain intensity; changes during treatment; from baseline to 6 months follow-up). | Week-0 (baseline), week-3 (mid-point of the treatment), week-6 (end of treatment), week-12 (mid-term follow-up), 6-month (long-term follow-up).
  Since DASH has few questions related to pain, the Brief Pain Inventory (BPI), which is specific for assessing clinical pain, will also be added to assess changes during treatment.
  The BPI measures pain intensity on an 11-point numerical rating scale (0-10), according to it interference with sleep, mood, etc., during the last 24 hours (ICC >0.80). Only the 4 first questions, related to clinical pain, will be used.
Symptoms (shoulder disabilities; changes during treatment; from baseline to 6 months follow-up). | Week-0 (baseline), week-3 (mid-point of the treatment), week-6 (end of treatment), week-12 (mid-term follow-up), 6-month (long-term follow-up).
  Because DASH is non-specific for shoulder, the "Western Ontario Rotator Cuff (WORC)" index will be added to assess changes at shoulder disabilities throughout treatment.
  The WORC is a reliable and responsive (ICC=0.96; SRM=1.54; MDC=12 points; CID=13 points) questionnaire designed to measure health-related-quality-of-life of patients affected by RC injuries.

SECONDARY OUTCOMES:
Range of Motion | Week-0 (baseline), week-6 (end of treatment).
  Active full and pain free range of motion in shoulder elevation in the frontal (abduction) and sagittal (flexion) planes will be measured using a digital inclinometer.
Acromiohumeral distance | Week-0 (baseline), week-6 (end of treatment).
  Outcome measurements at rest and 60º of active abduction using an ultrasound scanner.
Maximal electromyographic (EMG) amplitude | Week-0 (baseline), week-6 (end of treatment).
  Maximal EMG amplitude of infraspinatus, anterior and middle deltoid during full-range shoulder flexion and abduction.
Mean peak EMG amplitude | Week-0 (baseline), week-6 (end of treatment).
  Mean peak EMG amplitude of infraspinatus, anterior and middle deltoid during full-range shoulder flexion and abduction.
Onset timing | Week-0 (baseline), week-6 (end of treatment).
  Measurements at scaption (functional movement) using a slapping-ball task.

OTHER OUTCOMES:
Global Rating of Change | Week-6 (end of treatment).
  Participants will be asked to evaluate the change in their condition since the first physiotherapy session.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Sébastien Roy, PT, PhD, Study Director — Center for Interdisciplinary Research in Rehabilitation and Social Integration (CIRRIS), CIUSSS-CN; Fábio C L de Oliveira, PT, MSc, Principal Investigator — Center for Interdisciplinary Research in Rehabilitation and Social Integration (CIRRIS), CIUSSS-CN
Locations (1):
- Center for Interdisciplinary Research in Rehabilitation and Social Integration Research (CIRRIS), Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Oliveira FCL, Pairot de Fontenay B, Bouyer LJ, Desmeules F, Roy JS. Kinesiotaping for the Rehabilitation of Rotator Cuff-Related Shoulder Pain: A Randomized Clinical Trial. Sports Health. 2021 Mar;13(2):161-172. doi: 10.1177/1941738120944254. Epub 2020 Sep 28. PMID 32986531
- [Derived] de Oliveira FCL, Pairot de Fontenay B, Bouyer LJ, Desmeules F, Roy JS. Effects of kinesiotaping added to a rehabilitation programme for patients with rotator cuff tendinopathy: protocol for a single-blind, randomised controlled trial addressing symptoms, functional limitations and underlying deficits. BMJ Open. 2017 Sep 24;7(9):e017951. doi: 10.1136/bmjopen-2017-017951. PMID 28947462